CLINICAL TRIAL: NCT03242317
Title: A Prospective Study to Evaluate the Raindrop Near Vision Inlay in Presbyopes Treated With Mitomycin C During Surgery and Extended Steroid After Surgery
Brief Title: A Prospective Study to Evaluate the Raindrop Near Vision Inlay With Mitomycin C
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fichte, Endl & Elmer Eyecare (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FEE17-001
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Mitomycin C + Raindrop Near Vision Inlay (Experimental): The surgical procedure includes a low dose, short duration MMC treatment on the exposed stromal bed of the non-dominant eye, before the unilateral implantation of the Raindrop Near Vision Inlay in Presbyopes.
  Interventions: Drug: Mitomycin C; Device: Raindrop Near Vision Inlay

INTERVENTIONS:
Drug: Mitomycin C — The surgical procedure includes a low dose, short duration MMC treatment on the exposed stromal bed of the non-dominant eye, before the unilateral implantation of the corneal inlay. This treatment is at a concentration of 0.2 mg/mL (0.02%) applied for 10 to 30 seconds on the stromal bed as well as the stromal side of the corneal flap or pocket.
Device: Raindrop Near Vision Inlay — The surgical procedure includes the unilateral implantation of the Raindrop Near Vision Inlay in the non-dominant eye for the improvement of uncorrected near vision.

SUMMARY:
The objective of this study is to evaluate the Raindrop® Near Vision Inlay for the improvement of near vision in presbyopes treated with low dose, short duration Mitomycin C (MMC) during surgery and an extended low dose steroid regimen after surgery.

DETAILED DESCRIPTION:
The surgical procedure includes a low dose, short duration MMC treatment on the exposed stromal bed of the non-dominant eye, before the unilateral implantation of the corneal inlay. This treatment is at a concentration of 0.2 mg/mL (0.02%) applied for 10 to 30 seconds on the stromal bed as well as the stromal side of the corneal flap or pocket. In the third month after surgical procedure, one-drop a day of low dose steroid will be continued for the duration of the 24-month follow-up period to maintain corneal health.

ELIGIBILITY:
Inclusion Criteria:

Patients require a near reading add from +1.5 to +2.5 D in the non-dominant eye.

Patients have a photopic pupil size of at least 3.0 mm in the non-dominant eye. Patients have a corneal thickness greater than or equal to 500 microns in the non-dominant eye.

Patients have corrected distance and near visual acuity of 20/25 or better in each eye.

Patients have distance corrected near visual acuity of 20/40 or worse in each eye.

Patients are willing and able to sign and understand a written Informed Consent Form prior to any study-specific procedures.

Patients are willing and able to return for scheduled follow-up examinations for 24 months after the corneal inlay surgery.

Exclusion Criteria:

Patients with prior ocular surgery. Patients with clinically significant dry eye (i.e., significant diffuse punctate staining with fluorescein and a tear breakup time less than 8 s) in either eye.

Patients with a planned corneal residual bed thickness that is less than 300 microns (corneal thickness - (intended ablation depth + intended flap thickness)).

Patients with macular pathology based on dilated fundus exam and/or optical coherence tomography (OCT) image.

Patients who would be co-managed by an ophthalmologist or optometrist who is not approved as a ReVision Optics investigator.

Patients with ocular pathology or disease (including pupil pathology such as fixated pupils) that might confound the outcome or increase the risk of adverse event.

Patients taking systemic or topical medications that might confound the outcome or increase the risk of adverse event. Patients taking isotretinoin or amiodarone hydrochloride and any other medication that affects the tear film or accommodation, including but not limited to, mydriatic, cycloplegic and mitotic agents, tricyclic, phenothiazines, benzodiazepines, and first generation antihistamines.

Patients with known sensitivity to any planned study medications. Patients with residual, recurrent, active or uncontrolled eyelid disease. Patients with significant corneal asymmetry or irregular topography. Patients with clinically significant anterior segment pathology. Patients with any corneal abnormality, including but not limited to, slit lamp findings for corneal staining Grade 3 or higher, recurrent corneal erosion or severe basement membrane disease, and pterygium extending onto the cornea.

Patients with ophthalmoscopic/topographic signs of keratoconus or those who are keratoconus suspect.

Patients with history of Herpes zoster or Herpes simplex keratitis. Patients with any progressive retinal disease or subjects with a history or evidence of retinal vascular occlusion and/or hypercoagulability, because of the risks associated with high pressures during suction application.

Patients with known history of steroid-responsive intraocular pressure increases, glaucoma, preoperative IOP > 21 mm Hg, or are otherwise suspected of having glaucoma.

Patients with amblyopia or strabismus or those who are at risk for developing strabismus postoperatively as determined by corneal light reflex and cover-uncover testing.

Patients with diabetic retinopathy, collagen, vascular, diagnosed autoimmune disease (e.g., lupus, rheumatoid arthritis, fibromylagia), immunodeficiency (e.g., HIV), connective tissue disease, or clinically significant atopic syndrome such as allergies or asthma.

Patients on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing.

Patients with any type of active cancer (ophthalmic or non-ophthalmic). Patients with uncontrolled infections of any kind. Patients who are pregnant, lactating, of child-bearing potential and not practicing a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

Patients who actively participate in contact sports (i.e., boxing, martial arts) where impacts to the face and eye are a normal occurrence.

Patients participating in any other ophthalmic or non-ophthalmic drug/device clinical trials during the time of this clinical investigation.

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity | 24 Months
  After the inlay procedure, patients will attain functional near visual acuity in the inlay eye and functional distance acuity binocularly.

SECONDARY OUTCOMES:
Incidence of Corneal Reaction | 24 Months
  Patients treated with low dose, short duration MMC intraoperatively, then an extended low dose steroid regimen will have minimal levels of corneal reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Endl, MD, Principal Investigator — Fichte, Endl & Elmer Eyecare
Locations (1):
- Fichte Endl & Elmer Eyecare, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: No